CLINICAL TRIAL: NCT00446667
Title: A Pilot Safety Study of Inhaled Dry Powder Mannitol in Acute Exacerbations of COPD
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Failed to recruit
Sponsor: Syntara (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPM-COPD-HIP-101b
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: COPD; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: mannitol

INTERVENTIONS:
Drug: mannitol — 400mg BD for 2 days

SUMMARY:
COPD is a major cause of ill health and death in Australia with 40,000 hospital admissions, and a national cost of $898,000,000 annually. The gold standard treatment of COPD is steroids for inflammation, antibiotics for infection and bronchodilators and oxygen for respiratory failure. However, associated mucus hypersecretion is responsible for much of the inflammation and infection. The use of pharmaceutical agents to assist in the early clearance of the retained mucus has been limited, primarily because of lack of demonstrated effect. There has been a recent development of interest in pursuing new therapies for improving mucociliary clearance and several studies have demonstrated that clinical outcomes can be improved when osmotic agents such as mannitol are added to standard treatments. The purpose of this study is to conduct a pilot safety study in patients with an acute exacerbation of COPD to determine if it is safe to administer inhaled mannitol for facilitating mucus clearance.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 > 35% predicted
* COPD
* Exacerbation
* Inpatient

Exclusion Criteria:

* Pneumonia
* CO2 retention

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
FEV1 | 2 days

SECONDARY OUTCOMES:
safety | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: David Barnes, MBBS FRACP, Principal Investigator — Royal Prince Alfred Hospital NSW Australia
Locations (2):
- Australia (2):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales